CLINICAL TRIAL: NCT04420091
Title: Effect of Cartidyss-based Dietary Supplement on Knee Joint Functionality and Discomfort in Adult Population
Brief Title: Hydrolyzed Fish Cartilage Effect on Knee Joint Functionality and Discomfort in Adult Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abyss Ingredients (Industry)
Collaborators: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CARTIDYSS
Record Dates: First submitted 2020-05-28; First posted 2020-06-09 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Knee Discomfort
Keywords: knee discomfort; hydrolyzed fish cartilage; food supplement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cartidyss (Experimental)
  Interventions: Dietary Supplement: Cartidyss

INTERVENTIONS:
Dietary Supplement: Cartidyss — Oral intake of two tablets of Cartidyss 500 mg, once daily in the morning, preferably during a meal, with water, during 3 months

SUMMARY:
This study is an exploratory, non-comparative, multi-centric trial in 30 free-living healthy male and female subjects with moderate knee joint discomfort and loss of functionality.

The objective of this trial is to determine whether oral administration of Cartidyss, a concentrated fish cartilage extract, can contribute to the improvement of knee joint functionality and discomfort in adult population

DETAILED DESCRIPTION:
30 patients will be enrolled during a 4-month period in 3 investigational sites and each patient will undergo 3 visits (V0: Inclusion visit at baseline, V1: Follow-Up Visit after 1 month ± 3 day and V2: End Visit after 3 months ± 5 days).

The primary objective of this trial is to determine whether oral administration of Cartidyss, a concentrated fish cartilage extract, can contribute to the improvement of knee joint functionality and discomfort in adult population, using a specific self-administered questionnaire. The secondary objectives of the study are to evaluate the effect of Cartidyss on knee function and pain at rest and while walking, with patient global assessment and quality of life at each time point. The tolerance, compliance, satisfaction, rate of responder to the supplementation and pain killer's consumption would be also evaluated as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age limits (see above)
* Body Mass Index BMI ≤ 35 kg/m2
* Knee discomfort score at rest over the last 24 hours on the most painful knee evaluated on VAS (0-100) ≥ 40 at baseline
* Able to follow the instructions of the study
* Having signed an informed consent

Exclusion Criteria:

* related to knee:

  * Recent trauma (< 1 month) of the knee responsible of the symptomatic knee;
  * Concurrent articular disease interfering with the evaluation of knee pain left to the Investigator's discretion
  * Prosthesis in the target knee
* related to treatments:

  * Analgesics to manage knee pain 24 hours before inclusion visit;
  * Corticosteroids injection in the target knee in the last month;
  * Hyaluronan injection in the target knee in the last 6 months;
  * Arthroscopy in the last 6 months
  * Oral corticotherapy ≥ 5mg/day (in Prednisolone equivalent) in the last 3 months;
  * Symptomatic slow-acting drugs for osteoarthritis (SYSADOA) or dietary supplement, i.e., curcuma extract, chondroitin, glucosamine, diacerein or avocado-soya unsaponifiables int he last 3 months
  * Contraindications to Cartidyss: hypersensitivity or allergy to the product components (fish)
  * Treatments based on strontium ranelate, bisphosphonates, selective estrogen-receptor modulator (SERM) and parathormone (PTH) in the last 12 months
* related to associated diseases :

  * Any severe, uncontrolled and limiting diseases left to the Investigator's discretion
  * Anticipated need for any surgical or other invasive procedure during the trial including prosthesis in the target knee
  * Anticipated need for any forbidden treatments during the trial
  * Swallowing disorder
  * Patient with widespread pain/depression (e.g. fibromyalgia)
* related to patients:

  * Close collaborators to the investigational team, the study coordinator or to the Sponsor
  * Currently participating or having participated in another therapeutic clinical trial in the last 3 months
  * Under guardianship or judicial protection
  * Pregnancy, breastfeeding, planned conception, or premenopausal women without effective contraception (pill, patch, ring, diaphragm, implant and intrauterine device), tubal ligation or hysterectomy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of Cartidyss on knee functionality and discomfort after 3 months of supplementation | 3 months (Day 0, Month 1 and Month 3)
  Changes from baseline to 3 months of Knee injury and Osteoarthritis Outcome Score (KOOS) global score using a specific self-administered questionnaire Variation of Knee injury and Osteoarthritis Outcome Score using a self-administered questionnaire. The KOOS outcome score is a 42-item self-administrated questionnaire comprising 5 subscales: Pain, Symptoms, Activities of Daily Living, Sports and Recreation function, and Quality Of Life. A separate score ranging from 0 to 100, where 100 represents the best result, will be calculated for each subscale. A global score will be calculated by summing the score of each subscale.

SECONDARY OUTCOMES:
Evaluate the effect of Cartidyss on knee function after 3 months of supplementation | 3 months (Day 0, Month 1 and Month 3)
  Changes from baseline to each time points of knee function using the KOOS questionnaire, a specific self-administered questionnaire Variation of Knee injury and Osteoarthritis Outcome Score. The KOOS outcome score is a 42-item self-administrated questionnaire comprising 5 subscales: Pain, Symptoms, Activities of Daily Living, Sports and Recreation function, and Quality Of Life. A separate score ranging from 0 to 100, where 100 represents the best result, will be calculated for each subscale. A global score will be calculated by summing the score of each subscale.
Evaluate the effect of Cartidyss on knee pain at rest and while walking after 3 months of supplementation | 3 months (Day 0, Month 1 and Month 3)
  Changes from baseline to each time points. Variation of Visual Analogue Scale for the mean knee pain at rest and while walking over the last month The pain Visual Analogue scale (VAS) is a continuous scale comprised of a horizontal line, usually 10 centimeters in length (0-100mm), anchored by 2 verbal descriptors, one for each symptom extreme.
Evaluate the effect of Cartidyss on patient global assessment after 3 months of supplementation | 3 months (Day 0, Month 1 and Month 3)
  Changes from baseline to each time points. Variation of Visual Analogue Scale for patient global assessment of disease activity The Visual Analogue Scale (VAS) is a continuous scale comprised of a horizontal line, usually 10 centimeters in length (0-100mm), anchored by one verbal descriptors for Global Assessment of disease activity.
Evaluate the effect of Cartidyss on quality of life after 3 months of supplementation | 3 months (Day 0, Month 1 and Month 3)
  Changes from baseline to each time points. A global score will be calculated in function of the answers of a Self-administered questionnaire (SF-36). The SF-36 is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Evaluate the tolerance of Cartidyss after 3 months of supplementation | Only Month 1 and Month 3
  Number of Adverse events (AE or Adverse Device Effect or Device Deficiency; will be coded in terms of System Organ Class (SOC) and Low Level Terms (LLT) using the last version of MedDRA) and drop offs
Evaluate the compliance of Cartidyss after 3 months of supplementation | Only Month 1 and Month 3
  Count the capsules in investigation kits brought back by the patient.
Evaluate the satisfaction of Cartidyss after 3 months of supplementation | Only Month 1 and Month 3
  Changes after supplementation. Self-administered questionnaire using a 5-Likert scale (extremely unsatisfied- unsatisfied- nor unsatisfied nor satisfied- satisfied- extremely satisfied) to evaluate the product.
Evaluate the pain killer's consumption during the 3 months of supplementation | Only Month 1 and Month 3
  Changes after supplementation. Count the number of consumed pain killer
Evaluate the rate of responder to the 3 months supplementation of Cartidyss | Only Month 1 and Month 3
  Responder rate to treatment defined as changes in knee pain and/or knee function and/or patients disease activity according to the Outcome Measures in Rheumatology (OMERACT) and the OsteoArthritis Research Society International (OARSI) criteria. Responder criteria for osteoarthritis clinical trials based on the questionnaires describe above.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Chapelle, MD, Principal Investigator — Centre Médical Chant d'Oiseau (WOLUWÉ-SAINT-PIERRE)
Locations (2):
- Belgium (2):
  - Centre medical Chant d'Oiseau, Woluwe-Saint-Pierre - Sint-Pieters-Woluwe, Brussels Capital
  - Hopital Princesse Paola, VIVALIA, Marche-en-Famenne

REFERENCES:
- [Derived] Yves H, Herman J, Uebelhoer M, Wauquier F, Boutin-Wittrant L, Donneau AF, Monseur J, Fotso VM, Duquenne M, Wagner M, Bouvret E, Costes B, Wittrant Y. Oral supplementation with fish cartilage hydrolysate in an adult population suffering from knee pain and function discomfort: results from an innovative approach combining an exploratory clinical study and an ex vivo clinical investigation. BMC Musculoskelet Disord. 2023 Sep 21;24(1):748. doi: 10.1186/s12891-023-06800-4. PMID 37735385